CLINICAL TRIAL: NCT02219165
Title: Efficacy of IntraVenous ImmunoGlobulins (IVIG) in Toxic Shock Syndromes (Staphylococcal and Streptococcal): a Paediatric Pilot Study.
Brief Title: Efficacy of IntraVenous ImmunoGlobulins in Toxic Shock Syndromes: a Paediatric Pilot Study
Acronym: IVIG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2013.841
Record Dates: First submitted 2014-08-06; First posted 2014-08-18 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Toxic Shock Syndrome
Keywords: Paediatrics; Toxic Shock Syndrome; Intravenous human immunoglobulin; feasibility
MeSH Terms: conditions — Shock, Septic | interventions — Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG 2 g/kg (Experimental): Intravenous human immunoglobulin Day 1: As soon as there is suspicion of TSS, randomisation will be performed in order for the study treatment to be administered within the 12h following PICU admission (or following the manifestation of the first signs of shock). Concurrently, the TSS antibiotherapy following Surviving Sepsis Campaign recommendations is given
  Interventions: Drug: Intravenous human immunoglobulin
- Albumin 4% (Placebo Comparator): Same study scheduling as the first arm. Only the study treatment given is different (albumin instead of IGIV)
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Intravenous human immunoglobulin — Single administration of IVIG 2 g/kg within the 12 hours following PICU admission (or following the manifestation of the first signs of shock). The bottles of IVIG used will contain 10 g of proteins in 100 ml of solution. Thus, to reach a concentration of 2 g/kg, will be administered 1 bottle per 5 kg of body weight (with a maximum of 14 bottles for 70 kg patients and over).
  Arms: IVIG 2 g/kg
Drug: Albumin — Single administration of albumin 4% within the 12 hours following PICU admission (or following the manifestation of the first signs of shock). The solution will be given at the same volume as IVIG (that is: 1 bottle / 5 kg of body weight).
  Arms: Albumin 4%

SUMMARY:
Staphylococcus aureus and Streptococcus pyogenes produce many virulence factors. Some of them are responsible for severe infections in humans. Superantigen toxins synthesized by S. aureus or by S. pyogenes, are responsible for toxic shock syndromes (TSS) which lethality can attain 25% in children with validated criteria of septic shock.

Previous studies, performed in vitro and in vivo in animals, have shown that Intravenous immunoglobulins [IVIG] contain antibodies [Ab] against these toxins and, when used at high concentration, IVIG are able to neutralize their toxicity. However, in all these studies, IVIG administration has been preventive and there is no reliable data demonstrating their therapeutic efficacy in vitro or in vivo in humans or in animals, once the disease is present.

The efficacy of IVIG is established in other pathologies for which the role of the superantigens [superAg] is suspected, like Kawasaki disease in children. The mechanism of action, although not perfectly known, involves at the same time a direct effect on superAg (Ag-Ab complex) and indirect effects like the neutralisation of superAg within the network of anti-idiotype Ab or the neutralisation of the T-cells receptors. Staphylococcal and streptococcal toxic shocks imply bacterial exotoxins that are superAg. It seems thus consistent to imagine a same type of treatment with IVIG. However, there is currently no evidence of the efficacy of IVIG in this indication. One of the explanations relies on the lack of statistical power of previous adult studies, which principal objective was to show a reduction of the mortality. Taking into account the low prevalence of TSS, it has been hard to recruit enough patients to have the required statistical power. Moreover, some works have been extracted from larger studies on septic shock and the definitions of the TSS were nor always very reliable. Lastly, if the investigators consider the definition of the TSS as mentioned by the " Centre for Disease Control " [CDC], for which any hypotension, even a simple orthostatic hypotension, serves the diagnosis of TSS as long as the other symptoms are present, it is obvious that many patients are likely to be recruited in a study although it is highly probable that their health will get better with a " standard " treatment. The definition of a " real " TSS can be refined, keeping the CDC criteria, but changing the hypotension criterion in a more accurate criterion as described in the " surviving sepsis campaign ", internationally accepted and based on norms adapted to the age for paediatric forms.

IVIG therapy is very expensive and TSS is not recognized as indication of IVIG according to their marketing authorization. The feasibility of a randomized controlled study with this treatment needs to be assessed as it would be hazardous to conduct a large prospective RCT without having first assessed this feasibility in terms of recruitment rates, consent rates or compliance rates. Inclusion, randomisation and collect of inform consent in the context of severe shock are challenging and require evaluation of feasibility. The sample size calculation of the large study on mortality required estimations of the event in the specific population of children with criteria of septic shock. Surrogates markers of outcome need to be better defined. For example it would be useful to determine the evolution of organ dysfunctions with and without IVIG treatment in this population.

Various organ failure scores, used upon admission and later on, have been validated in adults and in children. The absence of improvement of the Paediatric logistic organ dysfunction (Pelod) score over time is a good indicator of mortality in Paediatric intensive care unit (PICU). It could be used as surrogate marker to evaluate the efficacy of IVIG.

ELIGIBILITY:
Inclusion Criteria:

* 1 month <Age < 18 years
* Admitted to PICU, with a strong suspicion of staphylococcal or streptococcal infection (at least one of the following criteria):
* Diagnostic of TSS according to CDC (Centre for Disease Control) criteria or Group A streptococcus necrotizing fasciitis (positive streptest) or Varicella with infected lesions and erythroderma or positive streptest or Erythroderma in menstrual period or Pleuropneumopathy with erythroderma or positive streptest in pleural fluid or Erythroderma and biological fluid positive to type A streptococcus ou staphylococcus (articular, pericardial, bronchopulmonar, pharynx…)
* with shock resistant to fluid resuscitation defined as the presence, despite 40 ml/kg of fluid volume in 1 hour, of: hypotension (<5th percentile) or systolic arterial pressure < 2 SD for age or need for vasoactive drugs in order to maintain AP at a normal level (dopamine > 5µg/kg/min or dobutamine, adrenaline, noradrenaline, milrinone whatever the dose) or 2 signs of hypo perfusion among: metabolic acidosis with a base deficit > 5 lactate x 2 laboratory normal value diuresis < 0,5 ml/kg/h capillary refill time > 5 sec difference skin/central temperature > 3°C
* Consent to participation

Exclusion Criteria:

* First signs of shock appeared more than 24h ago
* Known hypersensitivity to one of the components (study treatment or placebo)
* Hypersensitivity to homologous immunoglobulins, specifically in very rare cases of Ig A deficit, when the patient has anti-IgA antibodies
* Known hyperprolinemia
* Immunodeficiency (acquired or not)
* Immunosuppressive drugs
* No health cover

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | up to 12 months
  Measured in overall and in the different centers (eligibility, recruitment, refusal, non-respect of the inclusion/non-inclusion criteria)
Compliance with the protocol design | up to 15 months
  timing of randomization, respect of randomization and the interventions, respect of the blinding)
Practical feasibility | up to 15 months
  time required for the Case Report Forms completion, length of the interventions, missing data, difficulties met
Financial feasibility | up to 15 months
  budget per patient, personnel required

SECONDARY OUTCOMES:
Evolution of organ failure score (PELOD 2) | Day 1, day 2 and day 5
Mortality | D 60
Measure of the Cumulative vasopressor index (CVI) . | (a) before treatment (day 1) and after treatment (day 2) and (b) over the 24h following drug administration
Adverse events (AE) and serious AE | Day 1, day 2, day 3, day 4, day 5, PICU discharge, day 60
Mechanism of superantigens (ancillary biological study: immune response: HLA-DR, Treg pool) | Day 1, day 3/5, day 60
In vivo mechanism of IVIG (ancillary biological study: Vbêta, Ig dosage) | Day 1, day 3/5, day 60
measure of lactate clearance | (a) before treatment (day 1) and after treatment (day 2) and (b) over the 24h following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Javouhey, Principal Investigator — Service de réanimation pédiatrique, Hôpital Femme Mère Enfant, Groupement Hospitalier Est, 59 Boulevard Pinel, 69677 BRON, FRANCE
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

REFERENCES:
- [Result] Portefaix A, Dhelens C, Recher M, Cour-Andlauer F, Naudin J, Mortamet G, Joram N, Tissieres P, Ginhoux T, Kassai B, Boutitie F, Maucort-Boulch D, Javouhey E. High-dose intravenous immunoglobulin versus albumin 4% in paediatric toxic shock syndrome: a randomised controlled feasibility study. Arch Dis Child. 2024 Aug 16;109(9):717-723. doi: 10.1136/archdischild-2022-325274. PMID 38360044